CLINICAL TRIAL: NCT05910476
Title: A Randomized comparaTive Study Of Rosuvastatin/Ezetimibe 20/10mg and Atorvastatin/Ezetimibe 40/10mg in Patients With Coronary Artery Drug eLuting stEnt Implantation Requiring High-dose stAtin/Ezetimibe combiNaTion Therapy: TOLERANT Trial
Brief Title: Comparative Study of Rosuvastatin/Ezetimib 20/10 mg and Atovastatin/Ezetimib 40/10 mg (TOLERANT Trial)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: dotter (Unknown)
Responsible Party: Principal Investigator, Deok-Kyu Cho, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9-2023-0008
Record Dates: First submitted 2023-03-31; First posted 2023-06-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Dyslipidemias
MeSH Terms: conditions — Coronary Artery Disease; Dyslipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rosuvastatin/ezetimibe 20/10mg (Active Comparator): rosuzet 10/20mg
  Interventions: Drug: a high dose of statin/ezetimib
- atorvastatin/ezetimibe 40/10mg (Active Comparator): NB zet 10/40mg
  Interventions: Drug: a high dose of statin/ezetimib

INTERVENTIONS:
Drug: a high dose of statin/ezetimib — In randomization, 100 patients will proceed with Rosuvastatin/Ezetimib 20/10 mg and 100 patients will proceed with Atovastatin/Ezetimib 40/10 mg.
  A new generation of drug elution stents can be inserted and later registered, and if the patient agrees to participate in the study, they are randomly assigned after stent implantation.

SUMMARY:
the investigators would like to compare the differences between roschvastin and atovastatin in patients who require high-dose statin/ejetimib to undergo a new generation of drug elution stent implantation for cardiovascular disease and maintain LDL cholesterol below 55 mg/dL.

DETAILED DESCRIPTION:
Death from vascular disease accounts for about one-third of all causes of death. Important regulatory factors in cardiovascular disease include dyslipidemia, high blood pressure, and diabetes, and keeping LDL cholesterol low among dyslipidemia levels, especially after cardiovascular stent treatment, is an essential factor to prevent another event in the future. Statin is currently the most widely used LDL cholesterol control drug with multifunctional effects such as controlling inflammatory reactions, controlling the movement and proliferation of vascular smooth muscle cells, and inhibiting the production of blood clots in addition to LDL cholesterol control.In addition, in several clinical studies, statins have shown many effects in primary and secondary prevention of cardiovascular disease, and several studies have been published that lower LDL cholesterol results in more benefits. Based on these findings, the 2016 European Heart Association (ESC), 2018 American Heart Association (ACC), and most recently changed 2022 Korean guidelines recommend controlling LDL cholesterol to <55mg/dL for patients with coronary artery disease. However, high-dose statins alone are still difficult to maintain for a long time due to increased liver levels, diabetes, and muscle pain, and recently, a drug that lowers LDL cholesterol has been developed in the small intestine called Ezetimib and is widely used in combination with statins in actual clinical trials. In fact, the RACING trial published in LANCET for domestic patients reported that the combination of moderate-intensity statins (Rosuvastatin 10mg) and ezetimib had fewer side effects for three years and better compliance, resulting in a better rate of maintaining LDL cholesterol at 70mg/dL or less than high-intensity statins alone. However, in this study, the rate at which LDL cholesterol remained below 55 mg/dL after one year was only 42% for moderate statins/esetimibe and 25% for high-intensity statins, and remained similar for three years. Therefore, high-intensity statins and ezetimibes may be essential treatments to reduce LDL cholesterol to less than 55 mg/dL and more than 50% under the current new guidelines. High-strength statins usually refer to more than 40 mg of atovastatin and 20 mg of Rosuvastatin, and drugs that combine ezetimibe with these high-strength statins are currently widely used to lower LDL cholesterol to 55 mg/dL or less if there are no special side effects in clinical practice, but research on compliance is very insufficient. This study aims to observe the rate of discontinuation or intolerance in patients taking Rosuvastatin/Ezetimib 20/10mg and Atovastatin/Ezetimib 40/10mg, with no previous comparison, RACING trial reported a 5% rate of discontinuation at rosuvastain 20mg administered, and atovatin/10mg/10mg. Referring to On the use of a pilot sample for sample size determination. the hospital conducts about 60 PCI cases a month, and about 1/5 of them are expected to be able to enroll 100 patients per group for about two years to conduct a total of 200 patients.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older
2. Patients who underwent a new generation of drug elution stent implantation for cardiovascular disease

Exclusion Criteria:

1. LDL cholesterol levels below 55 mg/dL without statin treatment
2. Serum AST/ALT with an acute liver disease within a month or a normal upper limit that is not continuously explained
3. Allergies or overreactions to statins
4. Estimated Dawn of Less than 1 Year
5. If it is determined that follow-up is not possible for more than one year
6. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of statins changed | 12 months
  Percentage of statins changed to discontinuation or intolerance (muscle pain, muscle efficiency, elevated liver level, etc.) within a year
Rate at which LDL cholesterol remains below 55 mg/dL | 12 months
  Rate at which LDL cholesterol remains below 55 mg/dL in all 1-year blood tests

SECONDARY OUTCOMES:
The rate at which LDL cholesterol is maintained at 55 mg/dL in the blood test after a month | 1 months
  The rate at which LDL cholesterol is maintained at 55 mg/dL in the blood test after a month
Cardiovascular death | 12 months
  Cardiovascular death
number of non-fatal myocardial infarction | 12 months
  number of non-fatal myocardial infarction
number of non-fatal stroke | 12 months
  number of non-fatal stroke
number of coronary artery re-perfusion | 12 months
  number of coronary artery re-perfusion
number of Newly developed diabetes or difficulty in controlling sugar | 12 months
  number of Newly developed diabetes or difficulty in controlling sugar
occurrence of statin-related muscle symptoms requiring therapeutic or dose changes | 12 months
  occurrence of statin-related muscle symptoms requiring therapeutic or dose changes
Increased muscle enzyme aberration | 12 months
  Increased muscle enzyme aberration (CPK > 4 x normal upper limit)
Elevated liver enzyme levels | 12 months
  Elevated liver enzyme levels (AST, ALT, or both ≥ 3 x normal upper bound)
Elevated serum creatine levels | 12 months
  Elevated serum creatine levels (from >50% baseline)
number of Major bleeding | 12 months
  number of Major bleeding
number of people who stopped taking the drug | 12 months
  number of people who stopped taking the drug

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, Study Director — Yonsei University
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea